CLINICAL TRIAL: NCT04814940
Title: Retrospective Analysis of Real-world Data From Medical Records on the Use of Gonadotropin for Infertility Treatment to Describe the Treatment Patterns and to Understand the Clinical Impact
Brief Title: Retrospective Analysis of Real-world Data From Medical Records on the Use of MENOPUR for Infertility Treatment
Status: Withdrawn | Type: Observational
Why Stopped: Based on company decision to close the project
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000395
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-06

CONDITIONS: Infertility, Female
Keywords: MENOPUR
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MENOPUR Cohort — Non-interventional
  All directions for medication usage were solely at the discretion of the investigator in accordance with their usual routine clinical practice and are assumed to be consistent with the national prescribing information of the medicinal product in the country in which the study take place.

SUMMARY:
The purpose of this retrospective observational study is to describe the treatment patterns with MENOPUR and to understand the clinical impact for patients that underwent infertility treatment under real-world setting.

The primary objective is to describe the treatment patterns for the general population and for selected patient profiles.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult females who underwent ART treatment with MENOPUR for ovarian stimulation in 2018

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Adult females who underwent assisted reproductive technologies (ART) treatment with MENOPUR for ovarian stimulation in 2018
Study Population: Adult women, fitting the inclusion/exclusion criteria, who were prescribed MENOPUR in 2018 at for controlled ovarian stimulation in a treatment of infertility with In Vitro Fertilisation (IVF) or Intra-Cytoplasmic Sperm Injection (ICSI) will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment duration with MENOPUR (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Duration of treatment (in days) with MENOPUR for complete patient population and subgroup of patients will be reported. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of MENOPUR stimulation start (complete patient population and subgroups analysis) | At the day of the first MENOPUR injection during the ovarian stimulation treatment (during 20 days) in 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of MENOPUR stimulation end (complete patient population and subgroups analysis) | At the day of the last MENOPUR injection during the ovarian stimulation treatment (during 20 days) in 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Starting dose of MENOPUR prescribed in IU (complete patient population and subgroups analysis) | From day 1 up to day 20 of MENOPUR stimulation during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Dose Adjustment of MENOPUR in IU (complete patient population and subgroups analysis) | From day 1 up to day 20 of MENOPUR stimulation during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Total dose of MENOPUR (complete patient population and subgroup analysis) | From day 1 up to day 20 of MENOPUR stimulation during 2018
  Defined as total dose of MENOPUR used during the treatment duration. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Addition of gonadotropin (s) in case of mixed ovarian stimulation treatment (complete patient population and subgroup analysis) | Up to the end of the ovarian stimulation treatment (up to 20 days) during 2018
  In case of mixed treatments with gonadotropin (s) at the discretion of the investigator, addition of gonadotropin (s) will be reported. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Mixed treatment duration with added gonadotropin (s) (complete patient population and subgroup analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  In case of mixed treatments with gonadotropin (s), total duration with added gonadotropin (s) will be reported. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of treatment with additional gonadotropin (s) start (complete patient population and subgroups analysis) | At the day of the first additional gonadotropin (s) injection during the ovarian stimulation treatment (during 20 days) in 2018
  The time point of the start of the stimulation is decided at the discretion of the investigator. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of treatment with additional gonadotropin (s) end (complete patient population and subgroups analysis) | At the day of the last additional gonadotropin (s) injection during the ovarian stimulation treatment (during 20 days) in 2018
  The time point of the end of the stimulation is decided at the discretion of the investigator. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Starting dose of added gonadotropin (s) (complete patient population and subgroup analysis) | At the day of the first added gonadotropin (s) injection during the ovarian stimulation treatment (during 20 days) in 2018
  In case of mixed treatments with gonadotropin (s), starting dose of added gonadotropin (s) will be reported. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Dose adjustment of added gonadotropin (s) (complete patient population and subgroup analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Total dose of additional gonadotropin (s) (complete patient population and subgroup analysis) | Treatment prescription day with additional gonadotropin (s) up to the end of stimulation treatment (up to 20 days) during 2018
  Defined as total dose of additional gonadotropin (s) used during the treatment duration. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Type of gonadotropin releasing hormone (GnRH) used for Lutenizing Hormone(LH) surge suppression (complete patient population and subgroups analysis) | At consultation visit where the LH surge suppression protocol is decided during 2018
  Defined as a choice between GnRH agonist and GnRH antagonist. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of LH surge suppression protocol start (complete patient population and subgroups analysis) | At the day of the first GnRH administration during the ovarian stimulation treatment (during 20 days) in 2018
  The time point of the start of LH surge suppression is decided at the discretion of the investigator. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Day of LH surge suppression protocol end (complete patient population and subgroups analysis) | At the day of the last GnRH administration during the ovarian stimulation treatment (during 20 days) in 2018
  The time point of the end of LH surge suppression is decided at the discretion of the investigator. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Total number of follicles >=12 millimeter (mm) at the end of stimulation (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Circulating levels of progesterone (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Circulating levels of estrogen (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Type of drug used for the triggering of follicle maturation (complete patient population and subgroups analysis) | At consultation visit where the triggering of follicle maturation is decided during 2018
  Decided at the discretion of the investigator. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Date of administration of human chorionic gonadotropin (hCG) and/or GnRH for follicle maturation (complete patient population and subgroups analysis) | At the day of administration during 2018
  Date when the investigator decides to trigger the final follicle maturation. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Endometrium description: endometrial thickness (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Endometrium description: triple line visible (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Endometrium description: poorly defined central line (complete patient population and subgroups analysis) | Up to end of the ovarian stimulation treatment (up to 20 days) during 2018
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Type of drug used for Luteal phase support (complete patient population and subgroups analysis) | From ovum pick-up (OPU) day up to the end of luteal phase support during 2018
  Decided at the discretion of the investigator between progesterone, oestrogen and hCG. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.

SECONDARY OUTCOMES:
Number of oocytes retrieved (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Number of fresh or frozen embryo transfer (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Quality and number of embryo(s) transferred in fresh and frozen cycles (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Total number of embryo(s) and total number of good-quality embryo (s) transferred will be reported. Embryo quality is defined at the discretion of the investigator according to their routine practice. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Pregnancy rate (complete patient population and subgroups analysis) | 2 weeks after embryo transfer
  Defined as positive pregnancy 2 weeks after embryo transfer. Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Live birth rate (complete patient population and subgroups analysis) | At delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Live birth parameter: gestation duration (complete patient population and subgroups analysis) | At delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Live birth parameter: gender (complete patient population and subgroups analysis) | At delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Live birth parameter: weight (complete patient population and subgroups analysis) | At delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Percentage of pregnancy loss (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Number of patients with cycle cancellation before and after the ovum pick-up (OPU) (complete patient population and subgroups analysis) | From treatment prescription day with MENOPUR (during 2018) up to the OPU day during 2018 and from the OPU day during 2018 up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Percentage of preventive measures for early ovarian hyper-stimulation syndrome (OHSS) (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Rate of OHSS occurence (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.
Rate of early and late OHSS (complete patient population and subgroups analysis) | Treatment prescription day with MENOPUR (during 2018) up to the delivery
  Subgroup analysis refers to subgroups of patients stratified by patient baseline characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Assuta Medical Center Ltd, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
U.S. National Library of Medicine | U.S. National Institutes of Health | U.S. Department of Health & Human Services